CLINICAL TRIAL: NCT00968955
Title: Effect of Local Infiltration Analgesia With Ropivacaine in Total Hip Arthroplasty: a Prospective, Randomized, Double-blind, Placebo-controlled Trail
Brief Title: Effect of Local Infiltration Analgesia in Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Troels Haxholdt Lunn, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H-2-2009-079; 2009-41-3785
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Post-operative Pain
Keywords: Postoperative acute pain; Total hip arthroplasty; Local infiltration analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local infiltration with ropivacaine (Active Comparator): Local infiltration with ropivacaine 0,2% (150 ML)
  Interventions: Drug: Ropivacaine
- Local infiltration with saline (Placebo Comparator): Local infiltration with saline (150 ML) (placebo)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Local infiltration with ropivacaine 0,2% (150 ML)

SUMMARY:
The purpose of the study is to compare the effects of per-operative local infiltration analgesia with ropivacaine 0,2 % (150 ML) versus placebo on acute postoperative pain intensity after total hip arthroplasty.

The hypothesis is that local infiltration analgesia reduces the acute postoperative pain intensity.

DETAILED DESCRIPTION:
In spite of being one of the last century's most successful surgical procedures in treatment of advanced osteoarthritis total hip arthroplasty is still associated with postoperative pain and delayed rehabilitation. We therefore decided to evaluate the effects of per-operative local infiltration analgesia with ropivacaine 0,2 % (150 ML) versus placebo on acute postoperative pain intensity in a well defined, multimodal, fast-track setup after hip arthroplasty. The technique is widely used as standard treatment in many European centers despite its limited evidence.

ELIGIBILITY:
Inclusion Criteria:

* Elective total hip arthroplasty
* Able to speak and understand danish
* Able to give informed consent

Exclusion Criteria:

* Alcohol or medical abuse
* Allergies to local anesthetics
* Age < 18 years
* Daily use of opioids or glucocorticoids
* Pregnancy or breastfeeding
* Opioid intolerance
* Obesity defined as BMI>40 kg/m2
* Diabetic neuropathy and rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores on the Visual Analog Scale (during walking) | up to 8 hours

SECONDARY OUTCOMES:
Additional analgetics measured as cumulated amount i mg | up to 8 hours
Time spend in hospital measured as nights after surgery | At discharge (mean 2-3 nights)
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 8 hours
Postoperative pain scores on the Visual Analog Scale (at rest) | up to 8 hour

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Hvidovre University Hospital, Copenhagen, Hvidover
  - Hørsholm Hospital, Hørsholm, Hørsholm